CLINICAL TRIAL: NCT03467698
Title: Investigating Transcranial Direct Current Stimulation (tDCS) in Accelerating Learning in a Healthy Older Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Sven Vanneste, Associate professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18-40
Record Dates: First submitted 2018-02-28; First posted 2018-03-16 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Associative Memory in Healthy Subjects
Keywords: Aging; Memory; Associative learning; transcranial direct current stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups: (1) active tDCS (2) Sham tDCS.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active tDCS (Experimental): active HD-tDCS will be administered
  Interventions: Device: Active tDCS
- Sham tDCS (Sham Comparator): sham HD-tDCS will be administered
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — Real stimulation
  Arms: Active tDCS
Device: Sham tDCS — Sham stimulation
  Arms: Sham tDCS

SUMMARY:
The overall objective of this study is to explore whether transcranial Direct Current Stimulation (tDCS) can accelerate associative learning and boost associative memory in healthy subjects.

DETAILED DESCRIPTION:
The overall objective of this study is to explore whether transcranial Direct Current Stimulation (tDCS) can accelerate associative learning and boost associative memory in healthy subjects.

The aim of this study is to investigate the effects of transcranial Direct Current Stimulation (tDCS) stimulation during a verbal paired-associate learning task to determine if tDCS may be used as a way to enhance brain plasticity during an associative memory task, and to accelerate learning and to optimize associative memory performance. We hypothesize that participants who receive tDCS stimulation will improve their associative memory performance.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 55 and 75
2. Currently not using any medication contradicting with tDCS
3. Native English speaker
4. Capable of understanding and signing an informed consent

Exclusion Criteria:

1. Acquainted with the Swahili language or culture
2. Severe disease
3. Mental illness
4. Cardiac history
5. History of severe head injuries
6. History of epileptic insults
7. Any implanted devices such as pace maker, neurostimulator
8. Pregnancy

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2022-09-17 (Actual); Study Completion 2022-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Vanneste, PhD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- University of Texas at Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luckey AM, McLeod SL, Robertson IH, To WT, Vanneste S. Greater Occipital Nerve Stimulation Boosts Associative Memory in Older Individuals: A Randomized Trial. Neurorehabil Neural Repair. 2020 Nov;34(11):1020-1029. doi: 10.1177/1545968320943573. Epub 2020 Sep 23. PMID 32964776

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.533 (5.58) | 64.667 (5.78) | 64.60 (5.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 11
  Male | 6 | 13 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 13 | 13 | 26
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: A Computerized Verbal Paired-associate Memory Task Will be Used to Assess Memory Performance.
Description: Memory performance scores recorded in the computerized verbal paired-associate memory test during each visit will be compared between the two groups (active tDCS and sham tDCS).
Time Frame: Memory performance changes will be assessed in two different visits. First assessment (baseline) on visit 1 (learning), then one-week after during visit 2 (memory)
Measure: Mean (Standard Error); unit: percentage of words learned/remembered
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 15 | 15
percentage of words learned/remembered
  Visit 2 - memory | 38.036 (4.458) | 24.65 (3.458)
  Visit 1 - learning | 52.93 (25.87) | 58.93 (24.88)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2016-01-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT03467698/Prot_001.pdf